CLINICAL TRIAL: NCT06455943
Title: Evaluation of Thriving, Substance Use, Mental Health and Repeat Injury Among Participants in the THRIVE Program
Brief Title: Evaluation of Thriving, Substance Use, Mental Health, and Repeat Injury Among Participants in the THRIVE Program
Status: Not yet recruiting | Type: Observational
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: THRIVE001
Record Dates: First submitted 2024-06-06; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Violence; Assault

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to determine the impact of a hospital-based violence intervention program on a person's capacity to thrive and recurrent intentional injury. The aims of this study are:

1. To evaluate the impact of the HVIP on building personal capacity of youth who have experienced non-fatal violent injuries to thrive using:

   * Established measure changes in positive psychology and clinical metrics
   * A qualitative interview using thematic content analysis
2. Plot the methodology proposed to measure the impact of THRIVE on subsequent injuries using administrative data sources

Participants will complete surveys, participate in a semi-structured interview, and have their rate of recurrent intentional injury tracked over time.

Researchers will compare the rates of intentional reinjury between participants in the THRIVE program and those who present at other hospitals with similar injuries to see if there is a difference in the rate of recurrent intentional injury a 1, 5, and 10 years.

ELIGIBILITY:
Inclusion Criteria:

* ages 14-29
* presentation with an injury due to violence (defined as a gun shot wound, stab wound, blunt or bodily force, inflicted by someone else)
* participant in the THRIVE Program

Exclusion Criteria:

* unable to consent due to language barrier or brain injury
* sexual assault
* child abuse
* self-inflicted injury
* residence >1 hour from Toronto city limits

Ages: 14 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Youth injured by interpersonal violence who present at the emergency department of Unity Health Toronto - St. Michael's Hospital will be offered the hospital-based violence intervention program called THRIVE. THRIVE case managers connect with youth and provide supports in-hospital and in the community following discharge, providing wrap-around care with a strengths-based approach.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2035-07-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the impact of the HVIP on building personal capacity of youth who have experienced non-fatal violent injuries to thrive. | July 2024 - December 2025
  To evaluate changes in thriving, substance use, and mental health, validated measures and qualitative measures will be used. Quantitative measures collected using validated instruments will provide objective measures of change over time; while context-specific and nuanced growth will be captured through a semi-structured interview.
To pilot the methodology proposed to measure the impact of THRIVE on subsequent injuries within 1 year using administrative data sources | March - Sept 2026
  After 1.5 years of enrolment in THRIVE, study participants will be deterministically linked. Linkage will provide a wealth of baseline characteristics (demographics, income/marginalization), injury characteristics (ICD-10 coding patterns which can be contrasted to THRIVE documentation), as well as the capacity to follow these linked patients administratively over time and identify subsequent ED presentations and admission across any hospital in Ontario.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Snider, MD, FRCPC, Principal Investigator — Unity Health Toronto

IPD SHARING:
Plan to Share IPD: No